CLINICAL TRIAL: NCT05743556
Title: Comparison of the Effect of HILT and TRT on Muscle Tone in Cervicobrachial Syndrome
Brief Title: The Comparison of Effectivity Therapy by HILT and TRT in Muscle Hypertonus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Cemusova, HILT, TRT
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Muscle Tone Abnormalities; Muscle Spasm
Keywords: muscle tone; HILT; TRT; scalene muscle; levator scapulae; trapezius muscle
MeSH Terms: conditions — Spasm

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HILT group (Experimental): Therapy of muscle hypertonus by Hight intensive laser applied on cervical muscles.
  Interventions: Device: HILT laserotherapy
- TRT group (Active Comparator): Muscle hypertonus of the cervical area treated by Target radio frequency current.
  Interventions: Device: TRT therapy
- Control group (No Intervention): Group of patients with muscle cervical hyper tone without any therapy.

INTERVENTIONS:
Device: HILT laserotherapy — application of high intensive laser therapy on cervical muscles
  Arms: HILT group
Device: TRT therapy — application of radiofrekvention therapy on cervical muscles
  Arms: TRT group

SUMMARY:
Comparing the effect of high-intensity laser therapy (HILT) and targeted radiofrequency therapy (TRT) on muscle tone in the cervical and thoracic regions. The research aims to determine the effectiveness of the effect of novel physical therapy on the change of muscle tone in the cervical and thoracic region. This is an intervention experiment applied to a group of 60 probands.

DETAILED DESCRIPTION:
Approximately 60 probands, aged 18-60 years, with no gender preference, will be recruited from patients of an unnamed healthcare facility based on their voluntary participation while receiving a current indication for physiotherapy with a diagnosis of CB syndrome.

Subjects will be randomized into three groups. The first probands (n'20) will have HILT applied bilaterally to the mm. scalene, m.levator scapulae and m.trapezius pars descendens. The second group (n'20) will have TRT applied bilaterally to mm. scalene, m.levator scapulae and m.trapezius pars descendens. No physical therapy or physiotherapy will be used for the third group (n'20) for the duration of the study. Subjects will be examined and treated three times a week for a total of 6 times. The effect of each type of therapy will be demonstrated palpationally and subjectively using an analogue pain scale and an algometer. The obtained results will be further statistically processed.

ELIGIBILITY:
Inclusion Criteria:

* the presence of hypertonus in the mm.scalene, m.levator scapulae and m.trapezius pars descendens bilaterally
* tension demonstrated by palpation and subjective assessment of the patient on an analogue pain scale

Exclusion Criteria:

* Individuals with acute or infectious disease
* probands psychiatric diagnoses
* patients with cancers
* problems with skin integrity disorders
* other contraindications to the use of HILT and TRT

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
determine whether HILT causes a change in neck muscle tone after 6 applications | 15 minutes
  High- intensive laser therapy will be applied to m. scaleni, m. levator scapulae and m. trapezius. Before and after application, the degree of tenderness of the muscle will be determined using an algometer. This will be recorded in an Excel MS spreadsheet.
determine whether TRT causes a change in neck muscle tone after 6 applications | 15 minutes
  Radiofrekvention therapy will be applied to m. scaleni, m. levator scapulae and m. trapezius. Before and after application, the degree of tenderness of the muscle will be determined using an algometer. This will be recorded in an Excel MS spreadsheet.

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr., Study Director — Charles University Prague
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No